CLINICAL TRIAL: NCT02063477
Title: Effect of a French Maritim Pine Bark Extract Oligopin® on Blood Pressure: Double Blind, Crossover, Placebo-controlled Nutrition Intervention Trial
Brief Title: Effect of Oligopin® on Blood Pressure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Oligo_extract
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Product one (Placebo Comparator): 150 mg (maltodextrin)/day (75 mg maltodextrin included in 280 mg/gelule; 2 times/day: morning and evening) of Placebo plus Dietary Approaches to Stop Hypertension (DASH)
  Interventions: Dietary Supplement: Placebo
- Product two (Active Comparator): 150 mg Oligopin/day (75mg Oligopin included in 280mg/gelule; 2 times/day: morning and evening) of Oligopin® plus Dietary Approaches to Stop Hypertension (DASH)
  Interventions: Dietary Supplement: Oligopin®

INTERVENTIONS:
Dietary Supplement: Placebo — The placebo composition is for 1 gelule: 250 mg maltodextrin + 30 mg magnesium stearate; total weight: 280 mg/gelule
  Arms: Product one
Dietary Supplement: Oligopin® — Oligopin® PUR' expert (%) is a red brown powder extracted from the bark of the Maritime Pine (Pinus pinaster) with composition:
  - TOTAL POLYPHENOL CONTENT > 96
  1. MONOMERS + PHENOLIC ACIDS 30
  2. DIMERS >15
  3. OTHER OLIGOMERS 50
  PROCYANIDINS CONTENT (GPC) > 67
  The Oligopin composition is for 1 gelule: 75 mg Oligopin + 175 mg maltodextrine + 30 mg magnesium stearate: total weight: 280 mg/gelule
  Arms: Product two

SUMMARY:
The objective of the study is to evaluate the effect of consumption of a food supplement rich in procyanidins extracted from the bark of French pine, Oligopin®, on blood pressure of people with mild / moderate degree of hypertension. Furthermore, the effect Oligopin® consumption on markers involved in the development of hypertension, and endothelial function in key enzymes that regulate blood pressure, inflammation and oxidation are considered. Also, try to advance the understanding of the molecular mechanisms that regulate blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* early stages of hypertension (systolic BP ≥ 140 and ≤ 159 mm Hg) and/or diastolic BP: ≥ 90 and ≤ 99 mm Hg
* not receiving BP-lowering medication.
* obtained written informed consent before the initial screening visit.

Exclusion Criteria:

* Body Mass Index (BMI) > 30 kg/m2
* taking antihypertensive medications
* smoking
* pregnant or who intends to become pregnant
* wife in breastfeeding period
* persons with a self-reported history of clinical cardiovascular disease, cancer, chronic kidney disease (or a serum creatinine ≥ 1.7 mg/dL for men and ≥ 1.5 mg/dL for women) hypercholesterolemia (LDL-c ≤ 189 mg/dL, diabetes mellitus (or serum glucose ≥126 mg/dL), or consumption of more than 14 drinks of alcoholic beverages per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Differences detected on the time evolution of BP both in two arms of intervention | 5 weeks

SECONDARY OUTCOMES:
Anthropometric data (Weight, BMI, Waist circumference) | weeks 2, 5, 6, 9
Endothelial function (Laser-Doppler) | Weeks 2, 5, 6, 9
Biochemistry for on-going study control (Glucose, Total cholesterol levels, Creatinine, Albumine, Transaminases (GPT, GOT) | Week 1
- Biomarkers related with endothelial function (Endotheline-1, Nitrites (NO3), Nitrates (NO2)) - Biomarker related with blood pressure homeostasis (ACE activity) | Weeks 2, 5, 6, 9
- Biomarker related with inflammatory processes (High sensitive C Reactive Protein) - Biomarkers of antioxidant system (Oxidised- LDL levels, Reduced glutathione, Oxidised glutathione, Ratio Glutathione balance) | Weeks 2, 5, 6, 9

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M VALLS, PhD, Study Director — University Rovira i Virgili; Rosa SOLÀ, MD,PhD, Principal Investigator — Hospital Universitari Sant Joan, Universitat Rovira i Virgili, CTNS
Locations (1):
- Technological Center of Nutrition and Health (CTNS), Reus, Tarragona, Spain

REFERENCES:
- [Derived] Valls RM, Llaurado E, Fernandez-Castillejo S, Puiggros F, Sola R, Arola L, Pedret A. Effects of low molecular weight procyanidin rich extract from french maritime pine bark on cardiovascular disease risk factors in stage-1 hypertensive subjects: Randomized, double-blind, crossover, placebo-controlled intervention trial. Phytomedicine. 2016 Nov 15;23(12):1451-1461. doi: 10.1016/j.phymed.2016.08.007. Epub 2016 Aug 23. PMID 27765365